CLINICAL TRIAL: NCT02423837
Title: Prospective Multicenter Study: Bendamustine in Combination With Rituximab as a First-line Therapy Followed by Maintenance Therapy With Rituximab in Patients With Follicular Lymphoma
Brief Title: Bendamustine in Combination With Rituximab as a First-line Therapy Followed by Maintenance Therapy With Rituximab in Patients With Follicular Lymphoma
Acronym: BRiF
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Research Center for Hematology, Russia (Network)
Responsible Party: Principal Investigator, Elena N.Parovichnikova, MD, PhD, National Research Center for Hematology, Russia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FL-RUS-2013
Record Dates: First submitted 2014-04-14; First posted 2015-04-22 (Estimated); Last update posted 2015-04-22 (Estimated); Status verified 2015-04

CONDITIONS: Follicular Lymphoma
Keywords: follicular lymphoma; bendamustine; rituximab
MeSH Terms: conditions — Lymphoma, Follicular | interventions — Rituximab; Bendamustine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Rituximab, bendamustine

SUMMARY:
* To evaluate the efficacy of bendamustine in combination with rituximab as first line in patients with follicular lymphoma, 1-3A cytological type.
* To evaluate the safety, tolerability and feasibility of bendamustine in combination with rituximab as 1st line in patients with follicular lymphoma, 1-3A cytological type.
* To evaluate the impact of the regimen modification (bendamustine dose modification and/or extension of inter-cycle interval) into duration of complete and partial responses.
* To evaluate estimated treatment duration, reasons of treatment withdrawal.
* To evaluate the possibility of unification and standardization of therapy protocol BR (rituximab 375 mg/m2 on day 1 and bendamustine 90 mg/m2 on days 1-2).
* To evaluate factors affecting overall and progression-free survival.

DETAILED DESCRIPTION:
Protocol involves 6 courses of rituximab and bendamustine with 26 days interval between each course (one cycle continues 28 days). Control examination will be performed every two courses (28, 56, 84 days of treatment) and will include (physical examination, monitoring of clinical blood tests, biochemical blood tests, computed tomography, ultrasonography, in patients with gastrointestinal tract involvement - fibrogastroduodenoscopy and colonoscopy). Efficacy of therapeutic impact will be estimated as rates of complete remission, partial remission, stable disease or progression based on tumor size reduction comparing with pretreatment data and evaluated using computed tomography and expressed as a percentage. Patients with partial or complete remission or stable disease after 2 courses continue treatment. Patients with tumor progression excluded from issue. Patients which achieved a complete remission after 2 courses may end treatment after 4 courses.

Safety, tolerability and feasibility which implies hematologic and non-hematologic toxicity will be estimated using data of physical examination, monitoring of clinical blood tests, biochemical blood tests and bone marrow analyses (cytological, morphological and genetic tests).

ELIGIBILITY:
Inclusion Criteria:

* Patients with the diagnosis of follicular lymphoma confirmed by immunohistochemistry (IHC) analysis in the reference laboratory
* Written informed consent for the use of personal data approved by Independent Ethic Committee
* Men and women patients, 18-75 years old
* ECOG performance status ≤ 3
* No previous treatment with chemotherapy and/or radiation therapy of follicular lymphoma

Exclusion Criteria:

* The patient is participating in any clinical trials and/or receiving the experimental treatment.
* Transformation of follicular lymphoma to large cell lymphoma (for example, follicular lymphoma IIIB graduation, diffuse large B-cell lymphoma).
* Central nervous system involvement.
* The presence of a second malignancy within the last 5 years prior to the inclusion into the study except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer or prostate cancer.
* Clinically significant cardiovascular or cerebro-vascular disease in the past 6 months, such as acute myocardial infarction, unstable angina, significant ventricular arrhythmia, severe heart failure (NYNA class IV), stroke, or uncontrolled hypertension.
* Renal impairment (serum creatinine > 150 umol/L), except lymphoid infiltration of kidneys and tumor lysis syndrome.
* Liver failure (except leukemic/lymphoid organ infiltration), acute hepatitis (serum bilirubin > 2 x ULN, the activity of ALT and AST > 4 x ULN, prothrombin index < than 50%).
* Uncontrolled diabetes mellitus (serum glucose > 15 mmol/L)
* Sepsis (septicopyemic focuses, hemodynamic instability, inefficiency of antibacterial therapy) or acute infectious diseases.
* HIV, hepatitis B and C (including the absence of the Hbc and Hbs antibodies).
* Life-threatening bleeding, except of bleeding from the gastrointestinal tract caused by neoplastic process.
* Severe mental disorders (schizophrenia, major depressive syndrome and other productive symptoms).
* Physical failure requiring constant care, cachexia (total protein < 35 g/L).
* Known hypersensitivity to rituximab components.
* Known hypersensitivity to bendamustine components.
* Pregnant or currently breast-feeding woman
* Neutrophils count < 1500/mm3 and/or platelets count < 75000/mm3.
* Surgery prior 15 days before therapy initiation.
* In case of serious infectious complications relief, uncontrolled diabetes, hemorrhagic syndrome, hypertension patient may be included into the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2013-12; Primary Completion 2016-02 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
Efficacy (tumor size evaluation) | From date of randomization until ending of first line R-B therapy (up to 6 months)
  tumor size will be estimated using computed tomography, ultrasonography, fibragastroduodenoscopy and colonoscopy
hematologic and nonhematologic toxicity (changes in leukocytes and trombocytes count, hemoglobin concentration, biochemical blood tests, electrocardiography) | From date of randomization until ending of first line R-B therapy (up to 6 months)
  clinical blood tests, biochemical blood tests, electrocardiography

SECONDARY OUTCOMES:
complete or partial response rates | From date of randomization up to 90 months
  According to NCCN recomendations
hematologic and nonhematologic toxicity (clinical blood tests, biochemical blood tests, blood pressure measurement, pulse rate, electrocardiography) | From date of randomization up to 90 months
  clinical blood tests, biochemical blood tests, blood pressure measurement, pulse rate, electrocardiography
Dose reduction rate or interval elongation | From date of randomization up to 90 months
Number of patients which underwent full protocol | From date of randomization up to 90 months
lifespan without progression | From date of randomization up to 90 months

CONTACTS AND LOCATIONS:
Overall Officials: Sergey K Kravchenko, MD, PhD, Principal Investigator — National Research Center for Hematology
Locations (1):
- National Research Center for Hematology, Moscow, Russia